CLINICAL TRIAL: NCT04902690
Title: An Observation Monocentric Study to Analyse the Possible Neuroprotective Effect of Ocrelizumab Via VEGF Protein Expression in Relapsing Multiple Sclerosis Patients
Brief Title: The Possible Neuroprotective Effect of Ocrelizumab Via VEGF Protein Expression in Relapsing Multiple Sclerosis Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: VEGF Study
Record Dates: First submitted 2021-05-20; First posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Multiple Sclerosis Relapse
Keywords: Neuroprotective effect; Ocrelizumab; Multiple sclerosis; Vascular Endothelial Growth Factor
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood mononuclear cells (PBMCs) will be isolated from the blood of MS patients. Whole blood will be collected by venipuncture in Vacutainer tubes containing EDTA (BD). Samples will be collected without need for fasting.
  Whole blood will be collected at T0, T6 and T12.
  The protein content of all the samples will be determined by the Bradford protein assay method, employing bovine serum albumin as standard.
  RNA will be extracted from total PBMCs homogenates by using RNeasy Micro Plus Kit from Qiagen (Valencia, CA).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ocrelizumab (OCR) is a humanized anti-CD20 antibody approved for Relapsing Multiple Sclerosis (RMS) and Primary Progressive Multiple Sclerosis (PPMS), due to neuroprotective effects of partially unknown origin. While its mechanism of action is mainly thought to occur via B cell depletion, previous studies on rituximab, another anti-CD20 drug, showed that CD20 binding elicits several intracellular signalling pathways, also including Protein Kinase C (PKC) activation. Of interest, the β isoform of PKC is known to modulate, through the RNA-binding protein ELAV/HuR, the expression of Vascular Endothelial Growth Factor (VEGF), a signaling protein that has been suggested to play deleterious effects in the first phases of MS. Therefore, the hypothesis is that part of the neuroprotective effects exerted by OCR may also be due to the modulation of VEGF expression via PKCβ /HuR cascade. The primary objective is to evaluate the variation of the expression of VEGF (protein and mRNA) in Peripheral Blood Mononuclear Cells (PBMCs) induced by OCR therapy. No additional visits will be required outside of clinical practice. Additional laboratory testing (VEGF protein expression and PKCbeta/HuR cascade) will be performed on extra blood which will be taken during the routine blood exams.

This study is an observational, longitudinal, monocenter and single arm study, in patients with RMS who are newly prescribed with OCR as per clinical practice.

The study consists of the following visits as per clinical practice

* T0 visit: at the first dose of OCR, blood sample and clinical/radiological MS data will be collected.
* T6: after 6 months of OCR treatment, blood samples and clinical MS data will be collected.
* T12 visit: after 12 months of OCR treatment, blood samples and clinical MS data will be collected.

DETAILED DESCRIPTION:
Ocrelizumab (OCR) is a humanized monoclonal anti-CD20 antibody approved by the FDA in 2017 and by the European Medicines Agency in 2018 for treatment of adult patients with Relapsing Multiple Sclerosis (RMS). In addition, having shown neuroprotective effects, OCR is the first drug ever approved for early treatment of Primary Progressive MS (PPMS). Currently, OCR is thought to mostly act via the rapid depletion of the B cells expressing CD20. Additionally, this depletion most likely causes long-lasting changes in the profile of B cells, characterized by a reduction of their pro-inflammatory phenotype, as demonstrated with other anti-CD20 antibodies.

Of interest, previous studies on other anti-CD20 drugs, mainly rituximab, have shown that anti-CD20 agents also exert interesting effects on additional intracellular signaling pathways, such as those involving serine/threonine and tyrosine kinases, as well as c-myc. Considering the structural, pharmacokinetic and pharmacodynamic similarities between OCR and rituximab, it can be hypothesized that the efficacy of OCR in delaying disease progression and neuroprotection might also stem from such intracellular effects.

Among the various intracellular effects elicited by rituximab through the binding with CD20, stimulation of the Protein Kinase C (PKC) pathway is of potential significance. The term PKC encompasses a family of several serine/threonine protein kinases of which the isoform β has been implicated in pathological processes, such as diabetic retinopathy, via a specific PKCβ/HuR/Vascular Endothelial Growth Factor (VEGF) pathway (Amadio et al. 2010). Notably, HuR belongs to a family of RNA-binding proteins, named ELAV, which are able to influence virtually any aspect of the post-synthesis fate of the targeted transcripts, including VEGF.

VEGF is a signaling molecule involved in vital processes such as angiogenesis, endothelial proliferation and cellular response to hypoxia. The possible role of VEGF in MS pathogenesis and evolution has not been explored until recently, but mounting evidence points to the conclusion that VEGF might play a significant noxious role in the relapsing stage of MS, for instance by mediating an increase in blood-brain barrier (BBB) permeability, while playing a beneficial, neuroprotective role in the late, progressive stage of the disease. Of note, VEGF has a primary role in promoting vascular hyperpermeability, indeed via phosphorylation of endothelial tight junction proteins modulates their degradation, finally leading to BBB disruption. Further, it also regulates vessel growth and is chemotactic for monocytes and lymphocytes, promoting neuroinflammation.

Of interest, a significant increase in VEGF was observed in mice in the acute phase of murine MOG-induced MS, which correlates to the clinical score, and in sera of MS patients during clinical disease relapses.

Based on these considerations, it can be possible that OCR exerts an additional beneficial effect in MS therapy by modulating VEGF content.

With this project, we aim to explore the effects of OCR on intracellular signaling pathways by assessing VEGF expression in Peripheral Blood Mononuclear Cells (PBMCs) of RMS patients at the beginning of OCR therapy, as well as at 6 and 12 months of ongoing treatment.

In particular, ther purpose of the study is to focus on the pro-angiogenic VEGF-A 165, which seems the isoform mainly involved as mediator of inflammation and cellular immunity.

Further, the PKCβ/HuR cascade will be investigated in the same conditions. Secondly, disease activity during OCR treatment will be examined at every step, and also compared with VEGF and PKC levels.

The results will also possibly demonstrate a necessity of further determining the extent and significance of intracellular effects of anti-CD20 therapy in MS.

This study is an observational (phase 4) , longitudinal, monocenter and single arm study, in patients with RMS who are newly prescribed with OCR as per clinical practice.

The study consists of the following visits as per clinical practice:

* Baseline/start (T0): informed consent signature, inclusion/exclusion criteria verification, demographical characteristics, clinical medical history recording, concomitant therapies, neurological history recording (MS history), number of relapses from MS onset, neurological examination, the Expanded Disability Status Scale (EDSS), the Multiple Sclerosis Severity Score (MSSS), blood sample, ocrelizumab administration.
* T6: (after 6 months of OCR treatment) adverse events (including relapses), neurological examination, therapies changes, EDSS, MSSS, blood sample, ocrelizumab administration.
* T12 (after 12 months* of OCR treatment), adverse events (including relapses), neurological examination, therapies changes, EDSS, MSSS, blood sample, ocrelizumab administration.

ELIGIBILITY:
Inclusion criteria

* The participant must have a previous diagnosis of RMS in accordance with the 2017 revised McDonald criteria
* The participant must have been newly prescribed to OCR treatment according to clinical practice
* Absence of high dose of steroid treatment for at least 4 weeks
* The participant must be capable of giving signed informed consent.

Exclusion criteria

* Clinical MS relapse within four-week period prior to inclusion
* Pregnant or nursing (lactating) women.
* Chronic disease of the immune system, other than MS
* Active systemic bacterial, viral or fungal infections
* Allergy to OCR
* Already included in other interventional trials

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Patients with RMS, who are newly prescribed with OCR as per clinical practice, are enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2021-05-31 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
VEGF protein levels | Month 12 versus baseline (T0)
  To evaluate the expression of VEGF protein in PBMCs from patients with RMS

SECONDARY OUTCOMES:
VEGF protein levels | Month 6 versus baseline (T0)
  To evaluate the expression of VEGF protein in PBMCs from patients with RMS before and after OCR treatment.
VEGF mRNA levels | Change from baseline (T0) to Month 6 and Month 12
  To evaluate the expression of VEGF mRNA in PBMCs from patients with RMS before and after OCR treatment
PKCβ protein levels | Change from baseline (T0) to Month 6 and Month 12
  To evaluate the expression of PKCβ protein in PBMCs from patients with RMS before and after OCR treatment
PKCβ mRNA levels | Change from baseline (T0) to Month 6 and Month 12
  To evaluate the expression of PKCβ mRNA in PBMCs from patients with RMS before and after OCR treatment
Expanded Disability Status Scale (EDSS) | Change from baseline (T0) to Month 6 and Month 12
  To evaluate whether the expression of VEGF and PKCβ affects MS severity before and after OCR treatment.
  The Expanded Disability Status Scale (EDSS) is a method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability over time. The EDSS scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability.
Multiple Sclerosis Severity Score (MSSS) | Change from baseline (T0) to Month 6 and Month 12
  To evaluate whether the expression of VEGF and PKCβ affects MS severity before and after OCR treatment.
  The Multiple Sclerosis Severity Score (MSSS) relates scores on the Expanded Disability Status Scale (EDSS) to the distribution of disability in patients with comparable disease durations.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Bergamaschi, MD, Principal Investigator — IRCCS Mondino Foundation, Pavia

REFERENCES:
- [Background] Amadio M, Bucolo C, Leggio GM, Drago F, Govoni S, Pascale A. The PKCbeta/HuR/VEGF pathway in diabetic retinopathy. Biochem Pharmacol. 2010 Oct 15;80(8):1230-7. doi: 10.1016/j.bcp.2010.06.033. Epub 2010 Jul 1. PMID 20599775
- [Background] Di Girolamo F, D'Amato A, Lante I, Signore F, Muraca M, Putignani L. Farm animal serum proteomics and impact on human health. Int J Mol Sci. 2014 Sep 1;15(9):15396-411. doi: 10.3390/ijms150915396. PMID 25257521
- [Background] Girolamo F, Coppola C, Ribatti D, Trojano M. Angiogenesis in multiple sclerosis and experimental autoimmune encephalomyelitis. Acta Neuropathol Commun. 2014 Jul 22;2:84. doi: 10.1186/s40478-014-0084-z. PMID 25047180
- [Background] Hauser SL, Bar-Or A, Comi G, Giovannoni G, Hartung HP, Hemmer B, Lublin F, Montalban X, Rammohan KW, Selmaj K, Traboulsee A, Wolinsky JS, Arnold DL, Klingelschmitt G, Masterman D, Fontoura P, Belachew S, Chin P, Mairon N, Garren H, Kappos L; OPERA I and OPERA II Clinical Investigators. Ocrelizumab versus Interferon Beta-1a in Relapsing Multiple Sclerosis. N Engl J Med. 2017 Jan 19;376(3):221-234. doi: 10.1056/NEJMoa1601277. Epub 2016 Dec 21. PMID 28002679
- [Background] Li R, Rezk A, Miyazaki Y, Hilgenberg E, Touil H, Shen P, Moore CS, Michel L, Althekair F, Rajasekharan S, Gommerman JL, Prat A, Fillatreau S, Bar-Or A; Canadian B cells in MS Team. Proinflammatory GM-CSF-producing B cells in multiple sclerosis and B cell depletion therapy. Sci Transl Med. 2015 Oct 21;7(310):310ra166. doi: 10.1126/scitranslmed.aab4176. PMID 26491076
- [Background] Montalban X, Hauser SL, Kappos L, Arnold DL, Bar-Or A, Comi G, de Seze J, Giovannoni G, Hartung HP, Hemmer B, Lublin F, Rammohan KW, Selmaj K, Traboulsee A, Sauter A, Masterman D, Fontoura P, Belachew S, Garren H, Mairon N, Chin P, Wolinsky JS; ORATORIO Clinical Investigators. Ocrelizumab versus Placebo in Primary Progressive Multiple Sclerosis. N Engl J Med. 2017 Jan 19;376(3):209-220. doi: 10.1056/NEJMoa1606468. Epub 2016 Dec 21. PMID 28002688
- [Background] Moran EP, Wang Z, Chen J, Sapieha P, Smith LE, Ma JX. Neurovascular cross talk in diabetic retinopathy: Pathophysiological roles and therapeutic implications. Am J Physiol Heart Circ Physiol. 2016 Sep 1;311(3):H738-49. doi: 10.1152/ajpheart.00005.2016. Epub 2016 Jul 29. PMID 27473938
- [Background] Pascale A, Govoni S. The complex world of post-transcriptional mechanisms: is their deregulation a common link for diseases? Focus on ELAV-like RNA-binding proteins. Cell Mol Life Sci. 2012 Feb;69(4):501-17. doi: 10.1007/s00018-011-0810-7. Epub 2011 Sep 10. PMID 21909784
- [Background] Riley JK, Sliwkowski MX. CD20: a gene in search of a function. Semin Oncol. 2000 Dec;27(6 Suppl 12):17-24. PMID 11225995
- [Background] Roscoe WA, Welsh ME, Carter DE, Karlik SJ. VEGF and angiogenesis in acute and chronic MOG((35-55)) peptide induced EAE. J Neuroimmunol. 2009 Apr 30;209(1-2):6-15. doi: 10.1016/j.jneuroim.2009.01.009. Epub 2009 Feb 23. PMID 19233483
- [Background] Roxburgh RH, Seaman SR, Masterman T, Hensiek AE, Sawcer SJ, Vukusic S, Achiti I, Confavreux C, Coustans M, le Page E, Edan G, McDonnell GV, Hawkins S, Trojano M, Liguori M, Cocco E, Marrosu MG, Tesser F, Leone MA, Weber A, Zipp F, Miterski B, Epplen JT, Oturai A, Sorensen PS, Celius EG, Lara NT, Montalban X, Villoslada P, Silva AM, Marta M, Leite I, Dubois B, Rubio J, Butzkueven H, Kilpatrick T, Mycko MP, Selmaj KW, Rio ME, Sa M, Salemi G, Savettieri G, Hillert J, Compston DA. Multiple Sclerosis Severity Score: using disability and disease duration to rate disease severity. Neurology. 2005 Apr 12;64(7):1144-51. doi: 10.1212/01.WNL.0000156155.19270.F8. PMID 15824338
- [Background] Smith MR. Rituximab (monoclonal anti-CD20 antibody): mechanisms of action and resistance. Oncogene. 2003 Oct 20;22(47):7359-68. doi: 10.1038/sj.onc.1206939. PMID 14576843
- [Background] Theoharides TC, Konstantinidou AD. Corticotropin-releasing hormone and the blood-brain-barrier. Front Biosci. 2007 Jan 1;12:1615-28. doi: 10.2741/2174. PMID 17127408